CLINICAL TRIAL: NCT01095874
Title: Allogeneic Hematopoietic Stem Cell Transplantation Evaluation in High Risk Myelodysplasia: an Observational Non-interventional Study Comparing Outcome of Patients Aged From 50 to 70 Years With or Without Donor
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation Evaluation in High Risk Myelodysplasia: an Observational Non-interventional Study
Acronym: ONIalloMDS
Status: Completed | Type: Observational
Sponsor: Saint-Louis Hospital, Paris, France (Other)
Collaborators: Hospital Avicenne (Other); University Hospital, Grenoble (Other); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Principal Investigator, Marie Robin, Dr Marie Robin, Saint-Louis Hospital, Paris, France
Other Study IDs: AGRAAH 08-01
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Myelodysplasia
Keywords: myelodysplasia; allogeneic hematopoietic stem cell transplantation; Survival; Transplantation
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare outcome of high risk myelodysplasia patients aged from 50 to 70 years with or without HLA compatible (9 or 10 identities / 10) donor. High risk myelodysplasia includes IPSS intermediate 2 and high myelodysplasia and patients with sever thrombocytopenia. Patients are registered when they acquire risk factors.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 70 years
* For myelodysplasia other than CMML: patients can be included if they have at least one of these criteria:

  1. IPSSintermediate 1 and poor cytogenetics (complex, 3 or 7 abnormality);
  2. thrombopenia < 20x10ex9/L:
  3. IPSS intermediate 2 or high
* For CMML: patients can be included if they have at least one of these criteria:

  1. 2 of these criteria: hyperleucocytosis > 10x10exp9/L, splenomegaly>18cm, hemoglobin < 10gr/dl, platelet < 100x10ex9/L
  2. IPSS intermediate 2 or high

Exclusion Criteria:

* Patient not eligible for transplantation (including patients without donor)because of severe co-morbidity including:
* Renal failure with creatinine clearance < 30ml/min
* Cirrhosis or hepatic failure
* Respiratory disease with vital capacity < 30%
* Uncontrolled cardiac failure
* Uncontrolled neurological disease
* Poor performance status with karnofsky < or = 60%

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from 50 to 70 years with high risk myelodysplasia and eligible for transplantation
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2008-01; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
overall survival in patient with or without donor | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint-Louis, Paris, France